CLINICAL TRIAL: NCT02663843
Title: Comparison of 'Low Skill Fibreoptic Tracheal Intubation' Via I-gel® and Air-Q® Supraglottic Airway Devices in Patients With Simulated Difficult Airways.
Brief Title: Low Skill Fibreoptic Intubation I-gel vs Air-Q
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1601LSFOI
Record Dates: First submitted 2016-01-18; First posted 2016-01-26 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- i-gel airway (Experimental): I-gel inserted for the low skill fibreoptic intubation technique
  Interventions: Device: i-gel airway
- air-Q airway (Experimental): Air-Q inserted for the low skill fibreoptic intubation technique
  Interventions: Device: air-Q airway

INTERVENTIONS:
Device: i-gel airway — Fibreoptic intubation via i-gel airway device
  Arms: i-gel airway
Device: air-Q airway — Fibreoptic intubation via air-Q airway device
  Arms: air-Q airway

SUMMARY:
Tracheal intubation under general anaesthesia is the gold standard for securing the airway and for protecting the lungs against gastric aspiration. The conventional technique involves the use of a metal laryngoscope inserted into the mouth to create an air space, to allow insertion of an endotracheal tube.

Alternatively, an oral airway device (called a supraglottic device (SGD)) can be used for tracheal intubation. The SGD is first inserted. A fibrescope is inserted down the shaft of the SGD and into the trachea. This allows an endotracheal tube (previously pre-loaded onto the fibrescope) to be railroaded of the fibrescope and into the trachea. This technique is called 'low skill fibreoptic intubation' as the SGD acts as a guide for the fibrescope. Our study compares the performance of two SGD: i-gel and air-Q. The investigators will compare intubation success rate, insertion rate, and times for SGD insertion and intubation.

DETAILED DESCRIPTION:
The investigators are testing to see if fibreoptic intubation in patients via a supraglottic airway device i.e. 'low skill fibreoptic intubation' (LSFOI) is more successful via the i-gel® than in the air-Q®. Patients are those scheduled for elective surgery under general anaesthesia who would normally require tracheal intubation. The investigator's hypothesis is based on the results of the investigator's recent manikin study (CIRB 2014/2039). The investigators would like to see if this hypothesis translates to patients. It will also test secondary outcomes e.g. SGD insertion success rates and times, and intubation times. In the aforementioned manikin study, the air-Q® performed better with the SGD insertion rates and times. However, the i-gel® performed better with intubation success rates and times. The devices may perform different due to differences between the devices: design (shape, volume, length, aperture), material composition, and technique required for insertion and intubation.

24 adult patients undergoing elective surgery requiring general anaesthesia and endotracheal intubation in the major operating theater of Singapore General Hospital will be enrolled. The patient will then be randomised in equal proportions into two groups, either the air-Q® or i-gel®. Patients will undergo induction of general anaesthesia in a standardised fashion and in accordance with usual practice in the investigator's department of anaesthesia. Intubation will then proceed with the assigned airway device. Data collected will include successful endotracheal intubation, as evidenced by the presence of end tidal carbon dioxide on a capnograph. Time to intubation (from the initial handling of the airway device until successful intubation is confirmed with successful lung ventilation), the number of attempts required and the view achieved (according to the modified Cormack and Lehane scoring system) will also be recorded. Injuries to the lips, teeth or upper airway will be sought and documented by a blinded observer in the Post Anesthetic Care Unit.

A protocol will be provided to standardise the induction of general anaesthesia. This will involve the application of standard patient monitors, a period of pre-oxygenation, and administration of anaesthetic agents and muscle relaxants. If the patient desaturates to SpO2 < 94% during intubation, the intubation attempt via either the air-Q® or i-gel® will be abandoned and intubation will proceed using the conventional direct laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a physical status of American Society of Anesthesiologists (ASA) grade I/II and over 21 years old, having elective surgery, who require endotracheal intubation

Exclusion Criteria:

* ASA class III/IV
* Patients with history of previous difficult endotracheal intubation
* Patients with two or more predictors of difficult airway management (criteria 1-8, below)

  1. Airway masses
  2. Mallampati (oropharygneal space grading) III or IV
  3. Thyromental distance < 6.5cm
  4. Inter-incisor distance < 3 cm
  5. Head extension < 30 degrees
  6. Edentulous
  7. Large beard
  8. Obstructive sleep apnoea (OSA) or snorer
* Patients needing a rapid sequence induction
* Pregnant women

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Estimated); Study Completion 2017-06-01 (Estimated)

PRIMARY OUTCOMES:
Success of low skill fibreoptic intubation using the i-gel or air-Q airway devices measured end tidal carbon dioxide levels | 3 minutes
  Successful intubation indicated by normal end tidal carbon dioxide levels and trace

SECONDARY OUTCOMES:
Airway device insertion times | 3 minutes
  Time from picking up device to obtaining adequate canpography tracing
Low skill fibreoptic intubation times | 3 minutes
  Time from picking up fibrescope to obtaining adequate canpography tracing
Complication rate | Time of intubation and up to one day postoperative recovery period
  Complications due to airway and fiberscope insertion and use

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wong, Patrick, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospitals, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Lloyd LJ, Subash F, Wilkes AR, Hodzovic I. A comparison of fibreoptic-guided tracheal intubation through the Ambu (R) Aura-i , the intubating laryngeal mask airway and the i-gel : a manikin study. Anaesthesia. 2015 May;70(5):591-7. doi: 10.1111/anae.12988. Epub 2015 Jan 29. PMID 25631299
- [Background] Galgon RE, Schroeder KM, Han S, Andrei A, Joffe AM. The air-Q((R)) intubating laryngeal airway vs the LMA-ProSeal(TM) : a prospective, randomised trial of airway seal pressure. Anaesthesia. 2011 Dec;66(12):1093-100. doi: 10.1111/j.1365-2044.2011.06863.x. Epub 2011 Aug 22. PMID 21880031
- [Background] Moon HS, Lee JY, Chon JY, Lee H, Kim D. Air-Q(R)sp-assisted awake fiberoptic bronchoscopic intubation in a patient with Ludwig's angina. Korean J Anesthesiol. 2014 Dec;67(Suppl):S23-4. doi: 10.4097/kjae.2014.67.S.S23. No abstract available. PMID 25598892